CLINICAL TRIAL: NCT04881812
Title: A Randomized, Multi-center, Non-inferiority Clinical Trial on the Treatment of Residual Disease With Drug-Coated Balloon After Successful Recanalization and Limiting Stenting to the CTO Body Compared to Complete Stenting of the CTO Body and Adjacent Residual Disease.
Brief Title: Drug-Coated Balloon Coronary Angioplasty Versus Stenting for Treatment of Disease Adjacent to a Chronic Total Occlusion.
Acronym: Co-CTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Paul Knaapen, Principal Investigator, Professor of Interventional Cardiology, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VUmc_2020.0679
Record Dates: First submitted 2021-04-26; First posted 2021-05-11 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Drug-coated balloon; Drug-eluting stent; Randomized controlled trial; PCI
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: Patients with a CTO who are eligible for PCI will be randomized in a 1:1 ratio to additional DCB treatment or stenting of residual disease.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug-coated balloon (Experimental): Patients will receive stenting of the actual CTO body with additional DCB treatment of the residual disease of the coronary artery.
  Interventions: Device: Drug-Coated Balloons
- Drug-eluting stent (Active Comparator): Patients will receive complete stenting of the CTO body and residual disease of the coronary artery.
  Interventions: Device: Drug-Eluting-Stent

INTERVENTIONS:
Device: Drug-Coated Balloons — Percutaneous coronary intervention of residual disease adjacent to a chronic total occlusion with a paclitaxel drug-coated balloon (minimal stenting strategy).
  Arms: Drug-coated balloon
Device: Drug-Eluting-Stent — Percutaneous coronary intervention of the chronic total occlusion and residual coronary artery disease with an everolimus-eluting platinum chromium coronary stent (complete stenting strategy).
  Arms: Drug-eluting stent

SUMMARY:
This is an investigator-initiated, randomized, multi-center, non-inferiority clinical trial. Patients with a Chronic Total Occlusion who are eligible for PCI will be randomized to additional Drug-Coated-Balloon treatment or stenting of adjacent residual disease to the CTO body. The aim of this study is to investigate whether treatment with DCB is non-inferior to complete stenting of the CTO body.

DETAILED DESCRIPTION:
Rationale: Chronic total coronary occlusions (CTOs) are documented in approximately 16-18% of diagnostic coronary angiograms. New developments such as retrograde approach and dissection re-entry techniques have resulted in more widespread application of percutaneous coronary intervention (PCI) of CTOs, and this technique now serves as a viable alternative to optimal medical therapy alone or coronary artery bypass surgery. In general, PCI CTO is accompanied by extensive stenting of the coronary artery beyond the original occlusive segment itself. Unfortunately, stent length and diameter are directly related to poorer outcome, which is related to an increased rate of in-stent restenosis and thrombosis. An alternative to stenting is the application of drug-coated balloons (DCB). This strategy may prove beneficial, as it could significantly reduce stent length, among other things. However, data on the use of DCBs in the context of PCI CTO are currently lacking.

Objective: To investigate the value of DCB treatment in the residual disease of the coronary artery after successful recanalization and stenting of the actual CTO body as compared with complete stenting in a randomized fashion.

Study design: This is an investigator-initiated, randomized, single-blind (patients will be masked), multicenter, non-inferiority clinical trial.

Study population: 154 patients with a CTO eligible for PCI based on a formal local heart team decision will be screened for potential inclusion in the study.

Intervention: Patients with a CTO who are eligible for PCI will be randomized in a 1:1 ratio to additional DCB treatment or stenting of residual disease.

Main study parameters/endpoints: The primary endpoint is percentage diameter stenosis at 1-year follow-up as assessed by intravascular ultrasound (IVUS). Secondary invasive imaging objectives include minimal lumen diameter, late luminal loss, in-segment binary restenosis, and target vessel re-occlusion at 1-year follow-up. Secondary clinical objectives are evaluation of the occurrence of major adverse cardiac events (MACE) at 1-year follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group-relatedness: Participation in this study entails additional measurements, namely follow-up coronary angiography at 12 months, CCTA-scan at 12 months (if participating in substudy), and telephonic follow-up at 30 days and 12 months.

All patients included in the trial will have a clinical indication for percutaneous revascularization. Since there are no randomized controlled trials which advocate the use of either DES or DCB over one another in this setting, the risk of the PCI procedure will not be related to study participation. All patients will undergo coronary angiography after 1-year follow-up and will thus be exposed to the risks of invasive coronary angiography. Coronary angiography is characterized by a low complication rate (<0.5%). Repeat angiography also carries a low amount of radiation exposure. Patients participating in the CCTA substudy will be exposed to additional radiation. The ionized contrast agents used in both coronary angiography and CCTA substudy can be nephrotoxic and can elicit allergic reactions.

A DCB facilitated minimal stenting strategy for treatment of chronic total occlusions may significantly reduce stent length, number of used stents, as well as compression of the distal lumen with undersized stents. While DCB is expected to be non-inferior to DES regarding the in-segment diameter stenosis (primary endpoint), possible benefits may be observed in the secondary endpoints. Consequently, this trial could influence current guidelines on the application of DCBs in CTO procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical indication for revascularization of the CTO as determined by the local heart team (based on symptoms, documented ischemia, and viability)
* Successful recanalization of the CTO with residual disease adjacent to the initial lesion

Exclusion Criteria:

* Dissection affecting the flow (TIMI score<3), significant recoil (>30%) or coronary perforation after predilation
* Reference diameter of the vessel is <2.5 mm or >4.0 mm
* Bifurcation lesion requiring the stenting of the side branch
* Left main lesion
* Acute coronary syndrome
* Cardiogenic shock
* Severe kidney disease defined as an eGFR < 30 ml/min
* Pregnancy
* Life expectancy < 12 months
* Inability to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
In-segment diameter stenosis | 1 year
  The primary outcome is to investigate percentage diameter stenosis at 1-year follow-up as assessed by intravascular ultrasound (IVUS).

SECONDARY OUTCOMES:
Invasive | 1 year
  * Minimal lumen diameter (millimeters)
  * Late luminal loss (millimeters)
  * In-segment binary restenosis (>50%)
  * Target vessel re-occlusion (yes/no)
Clinical (MACE) | 1 year
  Major adverse cardiac events (MACE). MACE is composite endpoint of cardiac death, non-fatal myocardial infarction and ischemia driven target lesion revascularization (ID-TLR)
Clinical (angina) | At inclusion and 1-year follow-up
  Occurrence of angina pectoris according to the Canadian Cardiovascular Society Grading Scale (grade 1-4):
  1. Angina only during strenuous or prolonged physical activity;
  2. Slight limitation, with angina only during vigorous physical activity;
  3. Symptoms with everyday living activities, i.e. marked limitation;
  4. Inability to perform any activity without angina or angina at rest, i.e. severe limitation.

OTHER OUTCOMES:
Tertiary outcome | 1 year
  As measured in CCTA substudy:
  * Percent diameter stenosis (%)
  * In-segment binary restenosis (>50%)
  * Target vessel re-occlusion (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Knaapen, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - VUmc, Amsterdam, North Holland
  - Amsterdam Medical Center, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christopoulos G, Karmpaliotis D, Alaswad K, Yeh RW, Jaffer FA, Wyman RM, Lombardi WL, Menon RV, Grantham JA, Kandzari DE, Lembo N, Moses JW, Kirtane AJ, Parikh M, Green P, Finn M, Garcia S, Doing A, Patel M, Bahadorani J, Tarar MN, Christakopoulos GE, Thompson CA, Banerjee S, Brilakis ES. Application and outcomes of a hybrid approach to chronic total occlusion percutaneous coronary intervention in a contemporary multicenter US registry. Int J Cardiol. 2015 Nov 1;198:222-8. doi: 10.1016/j.ijcard.2015.06.093. Epub 2015 Jun 27. PMID 26189193
- [Background] Maeremans J, Walsh S, Knaapen P, Spratt JC, Avran A, Hanratty CG, Faurie B, Agostoni P, Bressollette E, Kayaert P, Bagnall AJ, Egred M, Smith D, Chase A, McEntegart MB, Smith WH, Harcombe A, Kelly P, Irving J, Smith EJ, Strange JW, Dens J. The Hybrid Algorithm for Treating Chronic Total Occlusions in Europe: The RECHARGE Registry. J Am Coll Cardiol. 2016 Nov 1;68(18):1958-1970. doi: 10.1016/j.jacc.2016.08.034. PMID 27788851
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] Fearon WF. Impact of drug-eluting stent length on outcomes less is more...more or less. JACC Cardiovasc Interv. 2010 Feb;3(2):189-90. doi: 10.1016/j.jcin.2009.12.006. No abstract available. PMID 20170876
- [Background] Suh J, Park DW, Lee JY, Jung IH, Lee SW, Kim YH, Lee CW, Cheong SS, Kim JJ, Park SW, Park SJ. The relationship and threshold of stent length with regard to risk of stent thrombosis after drug-eluting stent implantation. JACC Cardiovasc Interv. 2010 Apr;3(4):383-9. doi: 10.1016/j.jcin.2009.10.033. PMID 20398864
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO. 2018 ESC/EACTS Guidelines on myocardial revascularization. EuroIntervention. 2019 Feb 20;14(14):1435-1534. doi: 10.4244/EIJY19M01_01. No abstract available. PMID 30667361
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115
- [Background] Kleber FX, Rittger H, Bonaventura K, Zeymer U, Wohrle J, Jeger R, Levenson B, Mobius-Winkler S, Bruch L, Fischer D, Hengstenberg C, Porner T, Mathey D, Scheller B. Drug-coated balloons for treatment of coronary artery disease: updated recommendations from a consensus group. Clin Res Cardiol. 2013 Nov;102(11):785-97. doi: 10.1007/s00392-013-0609-7. Epub 2013 Aug 28. PMID 23982467
- [Derived] Somsen YBO, de Winter RW, Wu J, Hoek R, Sprengers RW, Verouden NJ, Claessen BEPM, Kleijn SA, Twisk JWR, Henriques JP, Spratt JC, Rissanen TT, McEntegart MB, Maehara A, Nap A, Knaapen P. Design and rationale of the drug-coated balloon coronary angioplasty versus stenting for treatment of disease adjacent to a chronic total occlusion (Co-CTO) trial. Am Heart J. 2025 Oct;288:65-76. doi: 10.1016/j.ahj.2025.03.023. Epub 2025 Apr 7. PMID 40204209